CLINICAL TRIAL: NCT00393614
Title: Levetiracetam Treatment of Children With Subclinical Sleep-Activated Epileptiform Activity (SSEA) - a Placebo Controlled Double-blind Cross-over-study
Brief Title: Levetiracetam Treatment of Children With Subclinical Sleep-Activated Epileptiform Activity (SSEA)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Ann-Sofie Eriksson, MD Phd, The National Centre for Epilepsy
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S06080; EudraCT number 2006-000795-32; SLV 200604331
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2008-02

CONDITIONS: Subclinical Sleep-Activated Epileptiform Activity; CSWS
Keywords: CSWS, interiktal epileptiform activity
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Care Provider, Investigator

INTERVENTIONS:
Drug: levetiracetam — 20 mg pr. kg a day

SUMMARY:
In clinical practice at the National centre for epilepsy (SSE) in Norway we see many children who have subclinical epileptiform activity in EEG that increases substantially during slow wave sleep (SSEA; subclinical sleep-activated epileptiform activity). They may or may not have seizures. Hence, according to the definition some children with SSEA do not suffer from epilepsy because they do not experience seizures. Many of these children have symptoms such as: attention deficit hyperactivity disorders (AD/HD), dyslectic problems, sleep problems, tantrums or autistic symptoms . We hypothesize that this subclinical epileptiform activity during slow sleep may act negatively on cognitive functions, language and behaviour in some children; even when the spike-wave discharges are less frequent than in CSWS (continuous spike-waves during slow sleep).

ELIGIBILITY:
Inclusion Criteria:

* Children 5-10 years
* IQ > 50

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
24 hour EEG | End of the study

SECONDARY OUTCOMES:
Neuro-psychological testing, | End of the study
Health related quality of life | End of the study
Behavioral problems | End of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Sofie Eriksson, MD Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Norway